CLINICAL TRIAL: NCT02619708
Title: Preoperative Immersive Patient Quality Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00028900
Record Dates: First submitted 2015-11-22; First posted 2015-12-02 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Patient-centered Outcomes Research; Surgery
Keywords: immersive preoperative experience

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Preoperative Experience (No Intervention): The preoperative visit will be performed, as it would be normally. Patients will be given a description of the preoperative experience, they will be told what to expect, they will be given brochures detailing what will happen on the day of the surgery, and will be given the opportunity to ask questions. Patients will fill out questionnaires immediately preoperatively on the day of the procedure, on the day after the procedure, and 30-days after the operation (only for patients undergoing surgery for degenerative spine disease).
- Immersive Preoperative Experience (Experimental): The preoperative visit will be performed, as it would be normally, with the only addition of a 5-minute video for the patients randomized to the intervention group. Patients will be given a few minutes to watch the video, and will have the chance to ask questions. The video will include a simulated patient encounter (with actors not real patients) showcasing the preoperative experience of the patient, including getting checked in, meeting the nurses, surgeons, and the anesthesiologists. Patients will fill out questionnaires immediately preoperatively on the day of the procedure, on the day after the procedure, and 30-days after the operation (only for patients undergoing surgery for degenerative spine disease).
  Interventions: Behavioral: Immersive Preoperative Experience

INTERVENTIONS:
Behavioral: Immersive Preoperative Experience — The video will include a simulated patient encounter (with actors not real patients) showcasing the preoperative experience of the patient, including getting checked in, meeting the nurses, surgeons, and the anesthesiologists. The technology used will allow the immersion of the patient in the preoperative environment. Patients will be able to look around and explore the spaces they will visit on the day of their operation.
  Arms: Immersive Preoperative Experience

SUMMARY:
In the current constantly changing healthcare landscape quality measurement has a central role. As the practice of medicine is shifting from authority to accountability, the quality of surgical interventions is under continuous scrutiny by patients, peers, payers, and policy makers. If done appropriately quality measurement can empower all members of the healthcare debate. There is increasing focus on patient satisfaction outcomes as quality indicators.

An important part of surgical outcomes is a patient's perception of the result of the intervention and overall experience in the preoperative setting. When assessing surgical outcomes, measuring patient satisfaction is necessary. A qualitative systematic review of patient satisfaction measures noted a scarcity of well-development quality improvement initiatives to improve patient satisfaction. Anxiety, a potent behavioral and psychological reaction, weighs heavily on a patient's perioperative experience and is exacerbated by preoperative concerns about underlying disease and impending anesthesia and surgery.

There are multiple stressors on the day of the surgery: unfamiliar environment, multiple forms to be signed, and multiple short encounters with new and unfamiliar personnel. These create confusion, increase baseline anxiety, and can negatively affect patient experience, and by extension surgical outcomes.

Increasing familiarity with this environment can help patients feel more informed about what matters most to them, and have more accurate expectations of possible benefits and harms of their options. This can potentially decrease overall anxiety, improve patient satisfaction, and decrease pain levels. With the current study investigators will have the following two specific aims:

Aim 1. To determine whether an immersive preoperative experience (video) is associated with decreased anxiety and improved patient experience during the perioperative phase.

Aim 2. To determine whether an immersive preoperative experience is associated with decreased stress, improved patient satisfaction, and decreased pain during the perioperative phase.

DETAILED DESCRIPTION:
The study will include patients scheduled to undergo neurosurgical interventions. Patients for whom surgical intervention is deemed necessary will be approached for participation in the study. After signing informed consent, they will be randomized to watch a video during their preoperative evaluation visit or have a regular standard of care evaluation during their preoperative visit. For the patients randomized to the intervention group, the preoperative visit will be performed, as it would be normally, with the only addition of a 5-minute video. Patients will be given a few minutes to watch the video, and will have the chance to ask questions. The remainder of the interaction between patient and provider will not be affected in any other way.

The video will include a simulated patient encounter (with actors not real patients) showcasing the preoperative experience of the patient, including getting checked in, meeting the nurses, surgeons, and the anesthesiologists. The technology used will allow the immersion of the patient in the preoperative environment. The hypothesis is that by introducing a way to familiarize the patients with the preoperative environment, investigators will have an impact on their anxiety about the operation and their satisfaction with the entire experience. Investigators hope this quality improvement initiative will change patient experiences for the better.

Patients will fill out questionnaires immediately preoperatively on the day of the procedure, on the day after the procedure, and 30-days after the operation (only for patients undergoing surgery for degenerative spine disease). The outcomes of interest will be stress level, pain level, and patient satisfaction level.

Preoperative, intraoperative, and postoperative variables will be analyzed using χ2 tests for categorical variables and the nonparametric Wilcoxon rank-sum test for continuous variables. Logistic regression will be performed, for each binary outcome. Linear regression will be performed, for each continuous outcome. The variable age will be tested separately as a continuous variable and a categorical variable (65-69 years, 70-74 years, 75-79 years, and ≥80 years) in multivariable logistic regression models. Other variables that will be included in the multivariable models include Charlson Comorbidity Index score, American Society of Anesthesiologists [ASA] score, APAIS score. Mixed effects methods will be used, with treating physician as a random effects variable, to account for clustering at the physician level.

Investigators intend to randomize 150 patients in 1:1 allocation to the video and conventional arms. We anticipate not being able to obtain the primary outcome on up to 10% of patients, leaving 135, or approximately 68 completers per arm. This yields just over 80% power at the usual 5% type 1 error rate to detect a difference between the two arms of one half (0.5) standard deviations in the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients undergoing elective neurosurgical procedures (brain, spine, peripheral nerve) under general anesthesia, for which a preoperative evaluation is undertaken

Exclusion Criteria:

* pediatric patients
* emergency procedures for which no preoperative visit has been scheduled
* patients that have undergone any prior operations, or had any exposure to the preoperative experience
* ability to complete a self-report questionnaire preoperatively and postoperatively
* cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2015-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
EVAN-G | Checked within 24 hours after the surgery
  A patient satisfaction score with 6 domains. The score ranges from 0-100 with higher scores representing higher satisfaction
APAIS | Checked immediately preoperatively on the day of the surgery
  A preoperative anxiety score with 6 domains. The anxiety score ranges from 4 to 20 and encompasses anxiety for the surgery and the anesthesia.

SECONDARY OUTCOMES:
Stress level | Checked immediately preoperatively on the day of the surgery
  On a scale of 0-100 with 0 being no stress and 100 being the worst stress in the patient's life. Visual Analog Scale
Pain level | Checked at 3 times: a) immediately preoperatively on the day of the surgery, b) within 24 hours after the surgery, and d) 30 days postoperatively
  On a scale of 0-100 with 0 being no pain and 100 being the worst pain in the patient's life. Will be checked for all patients at time points a) and b), and only for patients undergoing spinal operations for degenerative spine disease for time point c). Visual Analog Scale
Patient satisfaction level | Checked twice: a) immediately preoperatively on the day of the surgery, b) within 24 hours after the surgery
  On a scale of 0-100 with 0 being not satisfied and 100 being completely satisfied with the perioperative experience. Visual Analog Scale
Patient preparedness | Checked immediately preoperatively on the day of the surgery
  On a scale of 0-100 with 0 being not prepared and 100 being completely prepared for the perioperative experience. Visual Analog Scale

CONTACTS AND LOCATIONS:
Overall Officials: Kimon Bekelis, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Bekelis K, Calnan D, Simmons N, MacKenzie TA, Kakoulides G. Effect of an Immersive Preoperative Virtual Reality Experience on Patient Reported Outcomes: A Randomized Controlled Trial. Ann Surg. 2017 Jun;265(6):1068-1073. doi: 10.1097/SLA.0000000000002094. PMID 27906757